CLINICAL TRIAL: NCT03639402
Title: Protocol for Community-based Trial Among Nepalese Mothers With Young Children: Health Promotion Regarding Diet and Physical Activity
Brief Title: Cardiovascular Health Promotion Among Nepalese Mothers With Young Children (HARDIC Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HARDIC trial Nepal
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Diet Modification; Physical Activity; Health Behavior; Health Promotion
Keywords: Diet; Physical activity; Attitude; Knowledge; Practice; Cardiovascular disease; Mothers; Peer education
MeSH Terms: conditions — Motor Activity; Health Behavior; Behavior; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: one community is randomized as intervention arm, another community as control arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education classes (Experimental): Intervention consist of 2 rounds. Round 1: Locally selected mothers who have children 1-9 years old are trained by research team (peer mothers). Peer mothers conduct 4 education classes each for approximately 10 eligible mothers in their neighbourhood (fellow mothers).
  Round 2: After one month gap one meeting for recapitulation and feedback is conducted by research team for peer mothers. Similarly, peer mothers conduct one meeting with fellow mothers.
  Interventions: Behavioral: Health education classes
- No health education classes (No Intervention): Community is exposed to health-related information, which is provided by the regular health system of Nepal

INTERVENTIONS:
Behavioral: Health education classes — Community empowerment through involvement of local mothers (peer mothers) for dissemination of education regarding health diet and physical activity to others eligible mothers in the community (fellow mothers).
  Other Names: HARDIC trial
  Arms: Health education classes

SUMMARY:
Nutritional transition toward a high-fat and high-energy diet, decreasing physical activity level, and poor knowledge about cardiovascular health contribute to a rising burden of cardiovascular disease in low-income countries such as Nepal. Dietary and physical activity behaviors are formed early in life and influenced by family, particularly by mothers in the social context of Nepal. This is a community-based trial with health promotion intervention targeting mothers with young children regarding diet and physical activity. The intervention is designed based on the peer education approach. All mothers having children 1-9 years old living in study area are eligible for the participation in the trial. One of the two communities within the study site is randomly assigned as intervention arm and other as control arm. Selected local peer mothers from intervention arm are trained by research team regarding heart healthy diet and physical activity. In turn, peer mothers are conducting education classes to others local mothers living around them. Baseline and follow-up assessment of the intervention is covering mothers own knowledge, attitude and practice (KAP) regarding diet and physical activity and behavior of their children as perceived by mothers. Intention to treat analysis and per protocol analysis is used in analysis to detect significant differences between intervention and control group participants at baseline and follow-up. Difference in difference statistical analysis is chosen to evaluate real impact of the intervention in the community. Such community based intervention can further contribute to developing a policy that can be scaled-up to a national level.

DETAILED DESCRIPTION:
HARDIC project, includes needs assessment, development, and implementation of an intervention in the community, and also assesses impact. HARDIC trial is a community-based, randomized, controlled trial on diet and physical activity to promote heart health.

The studies is Jhaukhel-Duwakot Health Demographic Surveillance site (JD-HDSS), which consists of two villages-Jhaukhel and Duwakot-in the mid-hills of the Bhaktapur district, 13 kilometers outside Kathmandu, the capital of Nepal.

Baseline assesment to explore mothers' KAP regarding diet and physical activity is planned before intervention. Applying randomization (lottery method) Duwakot community is selected as intervention arm and Jhaukhel as control arm. Each community in Nepal is divided into nine administrative clusters (wards). To minimize contamination bias, the investigators selected five wards in Duwakot that did not border the control arm. The control arm includes all nine wards in Jhaukhel. HARDIC intervention is based on the concept of peer education for which 55 local peer mother from different wards of intervention arm are recruited with help of local female community health volunteers.

The intervention consists of two rounds. Selected peer mothers are divided into two groups and are trained by research team for 4 hours per day for 6 consecutive days. Training consists of interactive lectures, practical and demonstration sessions, discussions, group activities, practice sessions, and assignments. The peer mothers learn about communication skills and practiced using learning materials such as flipcharts. Additionally, home assignments for the 1-month gap between Rounds 1 and 2 is planned.

By the end of the training period, all peer mothers suppose to interact with neighbouring eligible mothers regarding the objectives of the intervention and accumulate a list of approximately 10 fellow mothers who are willing to participate in the intervention (educational classes given by peer mothers).

With the help of supervisors, peer mothers are preparing schedule for two 1-1.5-hour health education classes per week. Within 2 weeks after completing Round 1, each peer mother should conduct four health education classes for fellow mothers of their neighborhood. The health educational classes are based on the same modules that are used in the peer mothers' training and use the developed flipcharts, posters, and manuals for teaching purposes.

Round 2 is planned as providing recapitulation of the modules learned in Round 1 as well as discussion of the home assignments that peer mothers shall be given. Peer mothers follow same pattern when they teach fellow mothers.

Follow-up study is planned for both intervention and control arms in 3 months after completion of the intervention.

Mothers' KAP responses are scored and should be analyzed as continuous variables, calculated the median (IQR), and compared the intervention arm with control and KAP median (IQR) in the intervention arm at baseline and follow-up. Statistical Package for the Social Sciences (SPSS), version 23.0 (IBM, Armonk, New York, USA) shall be used for data management and analysis.

Actual impact of the intervention on mothers' KAP regarding diet and physical activity should be assessed using Difference in difference statistical approach from a linear regression model.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with children 1-9 years old

Exclusion Criteria:

* Mothers with hearing or mental disorders
* Mothers with mentally ill children or children whose health condition required a special diet and physical regimen
* Mothers who had lived in the community for only 2-3 months for seasonal work (eg, in brick kilns).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The aim of the project is to address diet and physical activity habits among young children to decrease possible risk of CVD in the future. In Nepal, mothers are mostly responsible for their family's food environment and also for shaping their children's lifestyle. Hence we enrolled mothers who have children 1-9 years old for the trial.
Enrollment: 1276 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 3 months
  Change in median of mothers' KAP scores regarding diet and physical activity

SECONDARY OUTCOMES:
Secondary outcome | 1 year
  Change in median of children's behavior scores regarding diet and physical activity as perceived by their mothers

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Oli, PhD, Principal Investigator — Kathmandu Medical College

IPD SHARING:
Plan to Share IPD: Yes
De- identified individual participant data will be made available. Data for baseline survey are available as a supplementary material in the publication in the PLOS One.
  Remaining data will be available after publishing the trial results.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Data will be available within 6 months after study completion
Access Criteria: Data access requests will be reviewed by external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.
URL: http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0200329